CLINICAL TRIAL: NCT04986722
Title: Cukurova University
Brief Title: Evaluation of Postoperative Nausea and Vomiting Incidence in Patients With Mastectomy Surgery According to Apfel Risk Scoring System
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hamide Sisman, Principal Investigator, Cukurova University
Other Study IDs: G-5097-2019
Record Dates: First submitted 2021-06-10; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To evaluate the symptoms of postoperative nausea and vomiting (PONV) in patients undergoing mastectomy with breast cancer according to the Apfel Risk Scoring System.

Materials and Methods: The descriptive and cross-sectional study was conducted between June 2020 and August 2020 in the surgical oncology department of a tertiary hospital. A total of 57 female patients who were scheduled for surgical treatment for breast cancer were included in the study. Data including demographic and clinical characteristics of the patients were recorded by face-to-face interview method. The incidence of PONV was evaluated using the Patient Evaluation Form and the Apfel Risk Scoring System.

DETAILED DESCRIPTION:
METHODOLOGY This descriptive, cross-sectional study was conducted at Department of Surgical Oncology of a tertiary care hospital between June 2020 and August 2020. The study centre has a 1,200-bed capacity and the surgical oncology clinic has a 30-bed capacity. A total of 57 women who were scheduled for elective mastectomy for breast cancer were included. Inclusion criteria were as follows: women aged ≥18 years, hospitalization 6 hours prior to surgery, American Society of Anesthesiologists (ASA) Class I-III, having no chronic pain or alcohol and/or substance abuse, having no cognitive impairment, no need for mechanical ventilation, having a confirmed diagnosis of breast cancer, and being scheduled for mastectomy. Prior to study, all patients were informed about the nature of the study and a written informed consent was obtained. The study protocol was approved by the institutional Non-Interventional Clinical Research Ethics Committee (No: 15.05.2020/99). The study was conducted in accordance with the principles of the Declaration of Helsinki.

Preoperative and postoperative data within 48 hours were collected via face-to-face interviews. The Patient Assessment Form, which was developed in accordance with the previous studies in the literature, was used to collect data including age and body mass index (BMI) pre- and postoperatively. For the postoperative evaluation, the four-item, simplified Apfel Risk Scoring System was used. It is a valid tool which assesses PONV and/or motion sickness, non-smoking status, and postoperative use of opioids. Accordingly, 0-1 indicate low, 2 indicate moderate, and ≥3-4 indicate high risk for PONV [12]. In our study, PONV was evaluated using the Patient Assessment Form at 0, 2, 4, 8, 24, and 48 hours as "Yes/No" scoring.

Statistical analysis was performed using the SPSS version 22.0 software (IBM Corp., Armonk, NY, USA). Descriptive data were expressed in mean ± standard deviation (SD), median (min-max) or number and frequency, where applicable. The chi-square test was used to evaluate relationship between categorical variables. The Mann-Whitney U test (Z table values) was performed to compare two independent groups which did not meet the normal distribution. The continuity correction and Fisher exact test were used to examine the relationship between two quantitative variables. The independent samples t-test (t table values) was used to compare two independent groups which met the normal distribution. A p value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer,
* Have female gender,
* Mastectomy planned

Exclusion Criteria:

* Having speech, comprehension and language barriers
* Who do not agree to participate in the study,
* Patients with male gender

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients scheduled for mastectomy
Study Population: - Patients diagnosed with breast cancer, female, scheduled for mastectomy, over 18 years of age and who agreed to participate in the study were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Apfel risk score before surgery | Preoperative 0-1 days
  Apfel Risk Scoring ; It is a tool in which the patient's previous postoperative nausea, vomiting and/or motion sickness history, non-smoking status, and postoperative opioid use are questioned to assess the patient's postoperative nausea and vomiting (PONV) risk score. The patient is evaluated with the Apfel Risk Score preoperatively. As a result of the evaluation, the patient is considered 0-1 point low risk, 2 points medium risk, and ≥3-4 points high risk for PONV.

SECONDARY OUTCOMES:
Evaluation of postoperative nausea and vomiting | Postoperative 0-2 days
  Using the Patient Evaluation Form, the patient's nausea and vomiting at 0, 2, 4, 8, 24 and 48 hours after the surgery was evaluated as "Yes/No" scoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.